CLINICAL TRIAL: NCT02568397
Title: Effect of LY3314814 on the Pharmacokinetics of Dabigatran in Healthy Subjects
Brief Title: A Drug-drug Interaction Study of Lanabecestat (LY3314814) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15997; I8D-MC-AZEE (Other: Eli Lilly and Company.)
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Healthy
MeSH Terms: interventions — lanabecestat; Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dabigatran Etexilate (Experimental): Single dose of dabigatran etexilate administered orally.
  Interventions: Drug: Dabigatran etexilate
- Lanabecestat and Dabigatran Etexilate (Experimental): Single dose of lanabecestat administered orally once daily on Days 3 to 21. Single doses of dabigatran etexilate administered orally on Days 16 and 20 during the lanabecestat dosing.
  Interventions: Drug: Lanabecestat; Drug: Dabigatran etexilate

INTERVENTIONS:
Drug: Lanabecestat — Administered orally
  Other Names: LY3314814; AZD3293
  Arms: Lanabecestat and Dabigatran Etexilate
Drug: Dabigatran etexilate — Administered orally

SUMMARY:
The purpose of this study is to learn about the effect of lanabecestat on how the body absorbs and processes dabigatran etexilate and how dabigatran etexilate affects lanabecestat when they are taken together. This study will last about 28 days and participants will be asked to take an lanabecestat tablet daily for 19 days and a dabigatran etexilate tablet on 3 occasions. Screening is required within 30 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

- Overtly healthy males and females

Exclusion Criteria:

* Eye abnormalities or disease
* History of vitiligo or any skin color disorder
* Have a history psychiatric or brain disease including seizures
* Have smoked within the last 3 months
* Are unwilling to avoid food and drinks containing grapefruit or Seville oranges for the duration of the study
* Have known allergies to dabigatran etexilate and related compounds

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10-31 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dabigatran Etexilate: Single dose of dabigatran etexilate administered orally on Day 1.
- LY3314814 + Dabigatran Etexilate: Single dose of LY3314814 administered orally once daily on Days 3 to 21. Single doses of dabigatran etexilate administered orally on Days 16 and 20 during the LY3314814 dosing
Period: Period 1
Arm/Group | Dabigatran Etexilate | LY3314814 + Dabigatran Etexilate
Started | 60 | 0
Received at Least 1 Dose of Study Drug | 60 | 0
Completed | 60 | 0
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Dabigatran Etexilate | LY3314814 + Dabigatran Etexilate
Started | 0 (A single oral dose of 150 mg dabigatran etexilate was administered on Day 1 of Period 1.) | 60 (Daily doses of 50 mg LY3314814 were administered daily on Days 3 to 21 of Period 2.)
Completed | 0 | 58
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Received at least one dose of study drug.
Groups:
- Overall: Overall study population
Arm/Group | Overall
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 31
  White | 25
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) : Maximum Concentration (Cmax) of Dabigatran
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, and 36 hours postdose
Population: All participants who received at least one dose of study drug and have evaluable pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Dabigatran Etexilate: Single dose of 150mg dabigatran etexilate administered orally on Day 1.
- LY3314814 and Dabigatran Etexilate Day 16: Single dose of LY3314814 administered orally once daily on Days 3 to 21. Concurrent single dose of dabigatran etexilate administered orally on day 16.
- LY3314814 and Dabigatran Etexilate Day 20: Single dose of LY3314814 administered orally once daily on Days 3 to 21.Single dose of dabigatran etexilate administered orally 4 hours after LY3314814 administration on Day 20.
Arm/Group | Dabigatran Etexilate | LY3314814 and Dabigatran Etexilate Day 16 | LY3314814 and Dabigatran Etexilate Day 20
Number analyzed (Participants) | 60 | 56 | 54
nanogram per milliliter (ng/mL) | 128 (69) | 148 (56) | 138 (46)

2. Primary Outcome: Pharmacokinetics: Area Under The Dabigatran Pharmacokinetic (PK) Concentration Versus Time Curve From Zero to Infinity (AUC[0-infinity)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, and 36 hours postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Dabigatran Etexilate | LY3314814 and Dabigatran Etexilate Day 16 | LY3314814 and Dabigatran Etexilate Day 20
Number analyzed (Participants) | 60 | 56 | 54
nanogram*hour per milliliter (ng*h/mL) | 1090 (61) | 1240 (53) | 1110 (44)

3. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Lanabecestat
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours postdose
Population: All participants who received one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- LY3314814 (AZD3293): 50 mg LY3314814 administered orally alone on Day 15.
Arm/Group | LY3314814 (AZD3293) | LY3314814 and Dabigatran Etexilate Day 16 | LY3314814 and Dabigatran Etexilate Day 20
Number analyzed (Participants) | 57 | 57 | 56
ng/mL | 342 (23) | 315 (21) | 331 (21)

4. Secondary Outcome: Pharmacokinetics: Area Under the Lanabecestat Pharmacokinetic (PK) Concentration Versus Time Curve During One Dosing Interval (24 Hours) (AUCtau)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose
Population: All participants who received one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- LY3314814 and Dabigatran Etexilate Day 20: Single dose of LY3314814 administered orally once daily on Days 3 to 21. Concurrent single dose of dabigatran etexilate administered orally on day 20.
Arm/Group | LY3314814 (AZD3293) | LY3314814 and Dabigatran Etexilate Day 16 | LY3314814 and Dabigatran Etexilate Day 20
Number analyzed (Participants) | 57 | 57 | 56
ng*h/mL | 3360 (25) | 3300 (26) | 3490 (24)

5. Secondary Outcome: Pharmacodynamics: Area Under the Effect Versus Time Curve (AUEC) of Thrombin Time
Time Frame: Days 1, 16 and 20: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, and 36 hours postdose
Population: All participants who received at least one dose of study drug and had evaluable Pharmacodynamic (PD) data.
Measure: Mean (Standard Deviation); unit: seconds*hour (s*h)
Groups:
- Dabigatran Extexilate Day 1: Single dose of 150 mg dabigatran etexilate administered orally on Day 1
Arm/Group | Dabigatran Extexilate Day 1 | LY3314814 and Dabigatran Etexilate Day 16 | LY3314814 and Dabigatran Etexilate Day 20
Number analyzed (Participants) | 57 | 55 | 49
seconds*hour (s*h) | 2080 (517) | 2170 (611) | 2030 (518)

6. Secondary Outcome: Pharmacodynamics: Ratio of Maximum Effect to Baseline Effect (ERmax) of Thrombin Time
Description: Ratio of maximum effect to baseline effect following administration of 150 mg dabigatran etexilate alone on Day 1, 50 mg LY3314814 and 150 mg dabigatran dosed concurrently on Day 16, and 50 mg LY3314814 and 150 mg dabigatran (dosed 4 hours later) on Day 20
Time Frame: Days 1, 16 and 20: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, and 36 hours postdose
Population: All participants who received at least one dose of study drug and had evaluable Pharmacodynamic (PD) data.
Measure: Median (Full Range); unit: ratio of maximum effect
Groups:
- Dabigatran Extexilate Day 1: Single dose of 150mg dabigatran etexilate administered orally on Day 1.
Arm/Group | Dabigatran Extexilate Day 1 | LY3314814 and Dabigatran Etexilate Day 16 | LY3314814 and Dabigatran Etexilate Day 20
Number analyzed (Participants) | 42 | 42 | 32
ratio of maximum effect | 7.10 [3.49 to 7.84] | 7.09 [1.06 to 7.84] | 7.00 [1.10 to 7.95]

ADVERSE EVENTS:
Groups:
- Dabigatran Etexilate: Single dose of 150mg dabigatran etexilate administered orally.
Arm/Group | Dabigatran Etexilate | LY3314814 (AZD3293) | LY3314814 and Dabigatran Etexilate Day 16 | LY3314814 and Dabigatran Etexilate Day 20
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 3/60 | 8/60 | 2/58 | 4/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dabigatran Etexilate (N=60) | LY3314814 (AZD3293) (N=60) | LY3314814 and Dabigatran Etexilate Day 16 (N=58) | LY3314814 and Dabigatran Etexilate Day 20 (N=58)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days